CLINICAL TRIAL: NCT06895980
Title: Effect of Periodontal Treatment on Metabolic Control in Patients with Type-2 Diabetes Mellitus Treated in the Cardiovascular Healt Program
Acronym: T2D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, MELISA VERA, Principal Investigator, Clinical Periodontist, Universidad de Chile, University of Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023/12; Gianina Cánnepa SPCH (Other: Periodontics Society of Chile)
Record Dates: First submitted 2025-03-13; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-09

CONDITIONS: Periodontitis Chronic Generalized Moderate; Periodontitis; Periodontal Disease; Diabetes Mellitus Type 2
Keywords: HbA1c; Periodontitis; Cardiovascular diseases; Diabetes mellitus; type 2 diabetes mellitus; scaling and root planing
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Longitudinal study of difference-in-difference
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with periodontitis and Diabetes Mellitus type 2 (Experimental): There will be a group of patients to intervene, who present periodontitis and Diabetes Mellitus type 2.
  Interventions: Procedure: Non-surgical periodontal treatment, glycated hemoglobin measurement and application of OHIP-14SP survey.

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment, glycated hemoglobin measurement and application of OHIP-14SP survey. — Non-surgical periodontal treatment will be performed, with periodontal maintenance therapy at 3, 6, 9 and 12 months, with measurement of glycated hemoglobin at each time and application of the OHIP-14SP oral health-related quality of life survey.

SUMMARY:
The objective of this clinical trial is to evaluate the effect of periodontal treatment on the reduction of glycated hemoglobin levels in adult patients with concurrent type 2 diabetes mellitus and periodontitis.

Non-surgical periodontal treatment and the application of a quality of life survey will be performed and then controls will be carried out for 1 year.

DETAILED DESCRIPTION:
The aim of this clinical trial is to evaluate the effect of periodontal treatment on the reduction of HbA1c levels in adult patients with type 2 diabetes mellitus who are users of the Cardiovascular Health Program and also to measure their quality of life by means of a survey OHIP-14sp.

Non-surgical periodontal treatment and subsequent follow-up of periodontal clinical parameters and HbA1c values at 3, 6, 9 and 12 months will be performed.

ELIGIBILITY:
Inclusion Criteria:

* 1a. Patients enrolled in the PSCV with a diagnosis of type 2 diabetes mellitus and who, in turn, have a glycated hemoglobin ≥ 7% (during the last 6 months).
* 1b. Patients with a diagnosis of periodontitis (≥ 2 non-adjacent teeth with detectable clinical interproximal attachment loss or, attachment loss ≥ 3mm with depth to probing ≥ 3mm on free faces of ≥ 2 teeth, where the attachment loss was not attributed to non-periodontal causes (Papapanou et al., 2018)).

Exclusion Criteria:

* 2a. Patients who have received periodontal treatment during the last year.
* 2b. Pregnancy/lactation, because they are under treatment under the Explicit Health Guarantee "Oral and Integral Health of Pregnant Women".
* 2c. Therapy with antibiotics and/or non-steroidal anti-inflammatory drugs (NSAIDs) in the last 6 months prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c (The glycated hemoglobin) | 13 months
  The glycated hemoglobin (HbA1c) is a blood test that measures the average blood glucose level over the past two to three months, expressed as a percentage. It is used to diagnose diabetes and prediabetes, and to monitor diabetes treatment.
  A higher percentage indicates poorer glycemic control. The value will be measured at the beginning of periodontal treatment and during maintenance therapy at 3, 6, 9 and 12 months.

SECONDARY OUTCOMES:
Patient self-reported quality of life. | 13 months
  Use of the OHIP-14 survey questionnaire that assesses people's quality of life in relation to their oral health.
  It is administered through questions that quantify the impact of oral disorders. It is based on 7 dimensions: physical pain, functional limitation, psychological discomfort, physical disability, psychological disability, and social disability.
  Scores range from 0 to 56 and are obtained by summing the ordinal values of the 14 items. Higher scores indicate a worse quality of life, and lower scores indicate a better quality of life.
  The Spanish version has been validated in older adults in Chile. We will apply the survey at the beginning of study and 12 months later.
Probing deep in periodontal evaluation | 13 months
  Probing depth is the distance between the gingival margin and the bottom of the periodontal pocket. It is measured in millimeters using a periodontal probe.
  It is measured at six points on each tooth. The probe is inserted parallel to the root surface in the periodontal pocket. It is moved around the gingival margin. In healthy areas, probing depth should not exceed 3 mm. Depths greater than 3.9 mm may indicate periodontal disease. We will administer this assessment at entry into the study and at 3, 6, 9, and 12 months.
Clinical attachment loss in periodontal evaluation | 13 months
  Clinical attachment loss is the difference between the position of the gum and the probing depth.
  It is measured at six points on each tooth using a periodontal probe. It is measured in millimeters.
  It is classified according to defined stages:
  Stage 1: 1 to 2 millimeters Stage 2: 2 to 3 millimeters Stages 3 and 4: 5 millimeters or more The assessment is performed at admission, and at 3, 6, 9, and 12 months.
bleeding of probing in periodontal evaluation | 13 months
  Bleeding on probing is a clinical parameter that indicates inflammation in the connective tissue of the gums.
  It is performed with a standardized periodontal probe. It is measured at six sites per tooth. It is a dichotomous variable, considered positive if bleeding occurs, or negative if no bleeding occurs.
  A value of less than 10% bleeding from all sites is considered periodontal stability.
  It will be assessed at admission and at 3, 6, 9, and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Melisa Vera, Specialist in periodontics, Principal Investigator — University of Chile
Locations (1):
- Universidad de Chile, Santiago, Providencia, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baeza M, Morales A, Cisterna C, Cavalla F, Jara G, Isamitt Y, Pino P, Gamonal J. Effect of periodontal treatment in patients with periodontitis and diabetes: systematic review and meta-analysis. J Appl Oral Sci. 2020 Jan 10;28:e20190248. doi: 10.1590/1678-7757-2019-0248. eCollection 2020. PMID 31939522
- [Background] Cobb CM. Clinical significance of non-surgical periodontal therapy: an evidence-based perspective of scaling and root planing. J Clin Periodontol. 2002 May;29 Suppl 2:6-16. PMID 12010523